CLINICAL TRIAL: NCT06120959
Title: Effect of Adding Pelvic Floor Exercises to the Stabilization Exercises in Treating Low Back Pain During Pregnancy: A Randomized Controlled Trial
Brief Title: Effect of Adding Pelvic Floor Exercises to the Stabilization Exercises in Treating Low Back Pain During Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Hany Ibrahiem, Master student at Department of Physical Therapy for Women's Health, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004252
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Related
Keywords: PELVIC FLOOR EXERCISES; STABILIZATION EXERCISES; LOW BACK PAIN; PREGNANCY
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group A (Active Comparator): They received exercise program in the form of Bridging, Seated Marching Twist, Quadruped pelvic tilts, Modified Side Plank, and Bird dog for 6 successive weeks.
  Interventions: Other: Stabilization exercise
- Study group B (Experimental): They received the same stabilization exercise program plus Pelvic floor exercise for 6 successive weeks.
  Interventions: Other: Stabilization exercise; Other: Pelvic floor exercise

INTERVENTIONS:
Other: Stabilization exercise — The exercise program included Bridging, Seated Marching Twist, Quadruped pelvic tilts, Modified Side Plank, and Bird dog for 6 successive weeks. .
Other: Pelvic floor exercise — The pelvic floor exercise protocol involved several steps. Prior to commencing the exercise, women were instructed to empty their bladders. The initial position for the woman was lying in a crook lying position. They were then guided to contract and hold their pelvic muscles for a duration of 5 to 6 seconds, followed by a relaxation period of 5 to 6 seconds. As the sessions progressed, patients were encouraged to perform the exercises in different positions: from a quadriped position, then sitting, followed by standing, and eventually while walking. Each session had a duration of 20 minutes, and the recommended frequency was three times a week for a span of 6 weeks. The repetitions were set at 10 to 15 per set, with two sets in total.
  Arms: Study group B

SUMMARY:
The purpose of the study is to know the effect of adding pelvic floor exercises to the stabilization exercises in treating low back pain during pregnancy.

DETAILED DESCRIPTION:
Low back pain (LBP) is a frequent condition in pregnancy, which may begin early, but the maximum pain out-put is typically found during the third trimester. (Adriana et al., 2020). LBP is pain or discomfort located between the 12th rib and the gluteal fold and PGP has been defined as 'pain experienced between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints' (Margie et al., 2018). LBP is a common health concern among women during pregnancy worldwide. The prevalence of LBP during pregnancy varies from and within sub regions. Moderate to severe disability associated with LBP is often a burden in pregnancy. The negative impact of LBP during pregnancy has implications on maternal quality of life and satisfaction with pregnancy. The duration of LBP in pregnancy correlates directly with the duration of absenteeism, physical dysfunction and poor work performance (Njoku et al., 2021).

The pelvic floor muscles (PFMs) are another component of the local stabilizing system, which in associated with deep abdominal and multifidus muscles play a critical role in lumbo-pelvic stability. Insufficiency can occur as a result of trauma, surgery, poor movement patterns, and childbirth. Previous studies reported that compared with healthy subjects, PFMs endurance time decreases in patients with pregnancy-related LBP (PRLBP). In addition, motor control of these muscles is altered in presence of sacroiliac join pain. Pregnancy can affect PFMs in several ways. The enhancement of hormonal level leads to muscle inhibition. Simultaneously, the growing of the uterus pushes pelvic organs downward and exert continuous strain on PFMs. Delivery itself changes the pelvic supportive system. These changes can impair PFMs function and load transferring in lumbo-pelvic area and lead to development of LBP. It was found that there is a synergistic relationship between local stabilizing muscles. Therefore, it could be supposed that a treatment program, which addresses local stabilizing muscles, can improve PFM function and decrease clinical symptoms in PRLBP (Zahra et al., 2018).

They were divided randomly into two equal groups using coin toss method;Group A (Control Group): consisted of 24 pregnant women with LBP and treated by routine treatment (Stabilization exercise) only 3 times per week for 6 successive weeks. Group B (Study Group): consisted of 24 pregnant women with LBP and treated by same program for group A and pelvic floor exercise only 3 times per week for 6 successive weeks.

ELIGIBILITY:
Inclusion Criteria:

* Their ages will range from 25-35 year.
* They will be at least in the 2nd trimester.
* Doesn't receive any treatment for her pregnancy-related low back pain.
* Low back pain with or without radiculopathy.
* Being in prenatal clinic follow up.

Exclusion Criteria:

* Previous pelvic floor muscle training.
* Previous pelvic / spine surgery.
* Structural anomaly.
* Urinary tract infection.
* Severe cardiovascular or metabolic disease.
* Twins or more.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 48 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The visual analogue scale (VAS) | 6 weeks
  The VAS is a quick and quite easy-to-use user-friendly instrument for rating pain. The VAS is a 10 cm line with descriptors at each end (from none to severe), along which respondents place a mark indicating their subjective pain. The score is measured as the distance of the mark from zero end of the line (Seyedehet.al.,2018). It was used to assess low back pain intensity for each woman in both groups before and after treatment.
Oswetry disability index (ODI) | 6 weeks
  The ODI is a reliable scale to detect improvement or worsening in most subjects with LBP. The questionnaire consists of 10 items of pain, lifting, self-care ability, the ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel. Each item is scored from 0-5, with higher values representing greater disability. The total score would be multiplied by 2 and expressed as a percentage. Zero means no physical disability and 100 mean the maximum disability (Seyedeh et al., 2018). It was used to assess functional disability for each woman in both groups before and after treatment.
Modified Schober Method | 6 weeks
  The Modified Schober Method was employed to assess lumbar flexion range of motion. The patient stood with specific spinal positions while the therapist marked anatomical points. A tape measure was used to quantify the flexion range of motion during forward bending

CONTACTS AND LOCATIONS:
Overall Officials: Dalia M. Kamel, Professor, Study Chair — Professor of physical therapy for women's health, Cairo University
Locations (1):
- Cairo University, Giza, Egypt